CLINICAL TRIAL: NCT02258464
Title: A Phase II Randomized, Double-blind, Placebo-controlled Trial of Radium-223 Dichloride Versus Placebo When Administered to Metastatic HER2 Negative Hormone Receptor Positive Breast Cancer Subjects With Bone Metastases Treated With Hormonal Treatment Background Therapy
Brief Title: Study of Radium-223 Dichloride Versus Placebo and Hormonal Treatment as Background Therapy in Subjects With Bone Predominant HER2 (Human Epidermal Growth Factor Receptor 2) Negative Hormone Receptor Positive Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to lower than expected recruitment since the start of study
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16298; 2014-002113-39 (EudraCT Number)
Record Dates: First submitted 2014-09-30; First posted 2014-10-07 (Estimated); Results first posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-07

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — radium Ra 223 dichloride; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Radium 223 dichloride (Experimental): Participants treated with a single hormonal agent as background therapy received 50 kBq/kg body weight (55 kBq/kg after implementation of National Institute of Standards and Technology [NIST] update) of Radium 223 dichloride intravenously for a maximum of 6 cycles at intervals of 4 weeks
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223); Other: Background hormonal therapy
- Placebo (Placebo Comparator): Participants treated with a single hormonal agent as background therapy received isotonic saline (0.9% sodium chloride solution for injection) intravenously for a maximum of 6 cycles at intervals of 4 weeks
  Interventions: Drug: Placebo (saline); Other: Background hormonal therapy

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — Up to 6 cycles of radium-223 dichloride 50kBq/kg body (55 kBq/kg after implementation of National Institute of Standards and Technology [NIST] update)
  Arms: Radium 223 dichloride
Drug: Placebo (saline) — Up to 6 cycles of saline injection
  Arms: Placebo
Other: Background hormonal therapy — Prescribed by PI and was provided as long as patient can tolerate treatment. It must be prescribed as per local label in country participating.

SUMMARY:
The objective of this study was to assess efficacy and safety of radium-223 dichloride in subjects with human epidermal growth factor receptor 2 negative (HER2 negative) hormone receptor positive breast cancer with bone metastases treated with hormonal treatment background therapy

ELIGIBILITY:
Inclusion Criteria:

* Documentation of histological or cytological confirmation of estrogen receptor positive (ER+) and HER2 negative adenocarcinoma of the breast must be available.
* Women (≥18 years of age) with metastatic breast cancer not amenable to curative treatment by surgery or radiotherapy.
* Documentation of menopausal status: post menopausal or premenopausal subjects are eligible.
* Subjects with bone dominant disease with at least 2 skeletal metastases identified at baseline by bone scintigraphy and confirmed by CT/magnetic resonance imaging (MRI). Presence of metastases in soft tissue (skin, subcutaneous, muscle, fat, lymph nodes)and/or visceral metastases is allowed.
* Measurable or non-measurable disease (but radiologically evaluable) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
* Subjects must have received at least one line of hormonal therapy in the metastatic setting
* Subjects who are eligible for further standard of care endocrine treatment.
* Subjects enrolled in the current study must start treatment with the single hormone agent either within 15 days prior to randomization or after randomization (before or simultaneously to the first injection of Ra-223/placebo).
* Subjects must have experienced no more than two skeletal-related events (SREs) prior to study entry defined as: Need for external beam radiotherapy (EBRT) tor bone, pathological bone fracture (excluding major trauma), spinal cord compression and/or orthopedic surgical procedure. Subjects with no prior SREs are not permitted.
* Subjects must be on therapy with bisphosphonate and denosumab. and are required to have been on such therapy for at least 1 month before start of study treatment.
* Adequate hematological, liver and kidney function.

Exclusion Criteria:

* Subjects with Inflammatory breast cancer.
* Subjects who have either received chemotherapy for metastatic disease or are considered by the treating investigator to be appropriate candidates for chemotherapy as current treatment for metastatic breast cancer are excluded. Chemotherapy administered for adjuvant/neo adjuvant disease is acceptable.
* Subjects with known or history of brain metastases or leptomeningeal disease: subjects with neurological symptoms must undergo a contrast CT scan or MRI of the brain within 28 days prior to randomization to exclude active brain metastasis. Imaging of the central nervous system (CNS) is otherwise not required.
* Known presence of osteonecrosis of jaw.
* Patients with immediately life-threatening visceral disease, for whom chemotherapy is the preferred treatment option.
* Lymphangitic carcinomatosis.
* Patients with ascites requiring paracentesis within 2 weeks prior to study entry (signature of informed consent) and during the screening period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (65):
- United States (11):
  - Bakersfield, California
  - La Jolla, California
  - Aurora, Colorado
  - New Haven, Connecticut
  - Cedar Rapids, Iowa
  - Annapolis, Maryland
  - Ann Arbor, Michigan
  - Pontiac, Michigan
  - St Louis, Missouri
  - Pittsburgh, Pennsylvania
  - Houston, Texas
- Austria (2):
  - Linz, Upper Austria
  - Innsbruck
- Canada (4):
  - Winnipeg, Manitoba
  - London, Ontario
  - Newmarket, Ontario
  - Toronto, Ontario
- Czechia (2):
  - Ostrava
  - Prague
- Denmark (2):
  - Copenhagen
  - Herlev
- Finland (2):
  - Helsinki
  - Tampere
- France (2):
  - Angers
  - Saint-Cloud
- Germany (3):
  - Tübingen, Baden-Wurttemberg
  - Bonn, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
- Kowloon, Hong Kong
- Ireland (2):
  - Cork
  - Dublin
- Israel (7):
  - Afula
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Ramat Gan
  - Tel Aviv
  - Ẕerifin
- Netherlands (2):
  - Nieuwegein
  - Zwolle
- Oslo, Norway
- Poland (3):
  - Bialystok
  - Gdynia
  - Warsaw
- Singapore, Singapore
- South Korea (4):
  - Busan
  - Daegu
  - Incheon
  - Seoul
- Spain (7):
  - L'Hospitalet de Llobregat, Barcelona
  - A Coruña
  - Barcelona
  - Madrid
  - Málaga
  - Seville
  - Zaragoza
- Aarau, Canton of Aargau, Switzerland
- Taipei, Taiwan
- United Kingdom (7):
  - Plymouth, Devon
  - Merseyside, Merseyside
  - Northwood, Middlesex
  - Nottingham, Nottinghamshire
  - Taunton, Somerset
  - Cottingham
  - Sheffield

REFERENCES:
- See also: Click here to find results for studies related to Bayer products. — http://clinicaltrials.bayer.com/
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 151 participants were screened at 69 active centers in 20 countries, the first participant first visit was on 02 Mar 2015 and last participant last visit was on 13 Aug 2019
Pre-assignment Details: Of the 151 screened participants, 99 participants (65.6%) completed screening and were assigned to treatment: 49 in the radium 223 dichloride and 50 in the placebo arm
Period: Overall Study
Arm/Group | Radium 223 Dichloride | Placebo
Started (Participants randomized in the study) | 49 | 50
Completed (Participants completed treatment of Radium 223/Placebo) | 32 | 25
Not Completed | 17 | 25
Not completed — Progressive disease (PD) | 9 | 17
Not completed — Study drug never administered | 1 | 1
Not completed — AE not related to clinical PD | 1 | 3
Not completed — Withdrawal by Subject | 5 | 4
Not completed — AE related to clinical PD | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intend-to-treat (ITT) analysis set: all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Radium 223 Dichloride | Placebo | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.08 (11.51) | 58.74 (11.97) | 57.92 (11.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 50 | 99
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 47 | 47 | 94
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 9 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 35 | 40 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Symptomatic Skeletal Event Free Survival (SSE-FS)
Description: Time from date of randomization to occurrence of one of the following, whichever happened earlier: 1) an on study SSE, which was defined as the use of external beam radiotherapy (EBRT) to relieve skeletal symptoms, the occurrence of new symptomatic pathological bone fractures (vertebral or nonvertebral), the occurrence of spinal cord compression, a tumor related orthopedic surgical intervention; or 2) death from any cause
Time Frame: Up to approximately 51 months
Population: Intent to treat analysis set: all randomized participants
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium 223 Dichloride | Placebo
Number analyzed (Participants) | 49 | 50
months | 30.1 (21.8) [21.8 to 43.0] | 18.4 (9.1) [9.1 to 28.2]
Statistical Analysis 1: Comparison: Radium 223 Dichloride vs Placebo; The null hypothesis that both treatment groups have the same SSE-FS distribution will be tested against the alternative hypothesis that the distribution of SSE-FS time in radium-223 dichloride is different from the placebo group; Test type: Other; p = 0.3339, Log Rank — The SSE-FS was compared using a stratified log-rank test with a 2-sided alpha of 0.2; Hazard Ratio (Radium 223/Placebo) = 0.745, 80% CI 2-sided [0.504 to 1.102]

2. Secondary Outcome: Overall Survival
Description: Time from randomization to death from any cause
Time Frame: Up to approximately 51 months
Population: Intent to treat analysis set: all randomized participants
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium 223 Dichloride | Placebo
Number analyzed (Participants) | 49 | 50
months | 43.0 [22.9 to NA] — NA: Value not estimated due to censored data | 32.4 [23.7 to NA] — NA: Value not estimated due to censored data
Statistical Analysis 1: Comparison: Radium 223 Dichloride vs Placebo; Test type: Other; p = 0.7259, Log Rank; Hazard ratio (Radium 223/Placebo) = 0.888, 80% CI 2-sided [0.576 to 1.370]

3. Secondary Outcome: Time to Opiate Use for Cancer Pain
Description: Interval from the date of randomization to the date of opiate use
Time Frame: Up to approximately 51 months
Population: Safety analysis set: all randomized participants who received at least one study drug administration (radium 223 dichloride or placebo)
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium 223 Dichloride | Placebo
Number analyzed (Participants) | 48 | 49
months | 21.3 [8.3 to NA] — NA: Value not estimated due to censored data | 20.2 [8.8 to NA] — NA: Value not estimated due to censored data
Statistical Analysis 1: Comparison: Radium 223 Dichloride vs Placebo; Test type: Other; p = 0.8785, Log Rank; Hazard ratio (Radium 223/Placebo) = 0.932, 80% CI 2-sided [0.513 to 1.693]

4. Secondary Outcome: Time to Pain Progression
Description: Time from randomization to the first date a participants (only in participants with baseline WPS ≤8) experiences pain progression based on worst pain score (WPS) ranging from 0 to 10 and analgesic use. Pain progression is defined as an increase of 2 or more points in the "Worst pain in 24 hours" score from baseline observed at 2 consecutive evaluations ≥4 weeks apart or an increase in pain management (IPM) with respect to baseline, whichever occurs first
Time Frame: Up to approximately 51 months
Population: as for outcome 3
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium 223 Dichloride | Placebo
Number analyzed (Participants) | 48 | 49
months | 14.8 [5.9 to 21.3] | 8.8 [3.7 to 14.3]
Statistical Analysis 1: Comparison: Radium 223 Dichloride vs Placebo; Test type: Other; p = 0.5240, Log Rank; Hazard ratio (Radium 223/Placebo) = 0.824, 80% CI 2-sided [0.556 to 1.220]

5. Secondary Outcome: Pain Improvement Rate
Description: The percentage of participants (baseline WPS>=2) with confirmed pain improvement at any time point. Confirmed pain improvement is defined as a 2 point decrease in worst pain score (WPS) from baseline over 2 consecutive assessment periods conducted at least 4 weeks apart
Time Frame: Up to approximately 51 months
Population: Participants in safety analysis set taken into account for this endpoint analysis
Measure: Number (80% Confidence Interval); unit: percentage of participants analyzed
Arm/Group | Radium 223 Dichloride | Placebo
Number analyzed (Participants) | 32 | 35
percentage of participants analyzed | 37.5 (25.9) [25.9 to 50.4] | 25.7 (16.2) [16.2 to 37.5]
Statistical Analysis 1: Comparison: Radium 223 Dichloride vs Placebo; Test type: Other; p = 0.345, Cochran-Mantel-Haenszel; Difference (Radium 223 - Placebo) % = 11.8, 80% CI 2-sided [-2.7 to 26.3]

6. Secondary Outcome: Time to Cytotoxic Chemotherapy
Description: Time from the date of randomization to the date of the first cytotoxic chemotherapy
Time Frame: Up to approximately 51 months
Population: Intent to treat analysis set: all randomized participants
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium 223 Dichloride | Placebo
Number analyzed (Participants) | 49 | 50
months | 16.0 (14.1) [14.1 to 22.4] | 17.3 (10.9) [10.9 to 27.6]
Statistical Analysis 1: Comparison: Radium 223 Dichloride vs Placebo; Test type: Other; p = 0.9128, Log Rank; Hazard ratio (Radium 223/Placebo) = 0.968, 80% CI 2-sided [0.657 to 1.425]

7. Secondary Outcome: Radiological Progression-free Survival (rPFS)
Description: Time from the date of randomization to the date of first radiological progression or death (if death occurs before progression)
Time Frame: Up to approximately 51 months
Population: Intent to treat analysis set: all randomized participants
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium 223 Dichloride | Placebo
Number analyzed (Participants) | 49 | 50
months | 8.1 (5.7) [5.7 to 10.6] | 5.8 (5.1) [5.1 to 7.9]
Statistical Analysis 1: Comparison: Radium 223 Dichloride vs Placebo; Test type: Other; p = 0.9227, Log Rank; Hazard ratio (Radium 223/Placebo) = 1.023, 80% CI 2-sided [0.753 to 1.391]

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Any event arising or worsening after the start of study drug administration until 30 days after the last study medication intake
Time Frame: Up to approximately 7 months
Population: Safety analysis set: all randomized subjects who received at least one dose of study medication (radium 223 dichloride or placebo)
Measure: Count of Participants; unit: Participants
Arm/Group | Radium 223 Dichloride | Placebo
Number analyzed (Participants) | 48 | 49
Participants
  Any TEAE | 46 | 46
  Radium 223/Placebo related TEAEs | 21 | 16

9. Secondary Outcome: Number of Participants With Post-treatment Adverse Events Including Additional Malignancies and Chemotherapy Related Adverse Events
Description: AEs related to the study drug, all occurrences of additional malignancies, febrile neutropenia and hemorrhage in subjects receiving chemotherapy, bone fractures and bone associated events (regardless of severity and relationship to study drug), and some symptoms needed for the characterization of an symptomatic skeletal event
Time Frame: From 30 days after the last dose of study treatment until the end of study, assessed up to approximately 44 months
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Radium 223 Dichloride | Placebo
Number analyzed (Participants) | 48 | 49
Participants
  Any post-treatment AE | 15 | 16
  Anaemia | 1 | 0
  Febrile neutropenia | 0 | 1
  Chest pain | 0 | 1
  Fibula fracture | 0 | 1
  Rib fracture | 0 | 1
  Tibia fracture | 0 | 1
  Traumatic fracture | 2 | 4
  Weight decreased | 0 | 1
  Arthralgia | 1 | 0
  Back pain | 4 | 0
  Bone pain | 2 | 3
  Muscle spasms | 1 | 0
  Musculoskeletal chest pain | 1 | 0
  Osteonecrosis of jaw | 1 | 0
  Pain in extremity | 1 | 1
  Pathological fracture | 5 | 4
  Spinal pain | 0 | 3
  Cauda equina syndrome | 0 | 1
  Paraesthesia | 0 | 1
  Spinal cord compression | 1 | 1
  Acute kidney injury | 0 | 1

ADVERSE EVENTS:
Time Frame: From the start of study drug administration until the end of study, assessed up to approximately 51 months
Description: Adverse events (AEs) included 1) any event arising or worsening after the start of study drug administration until 30 days after the last study medication intake 2) AEs related to study treatment reported beyond 30 days after study medication, all occurrences of additional malignancies, febrile neutropenia and hemorrhage in subjects receiving chemotherapy, bone fractures and bone associated events and and some symptoms needed for the characterization of an symptomatic skeletal event
Arm/Group | Radium 223 Dichloride | Placebo
All-Cause Mortality (participants affected / at risk) | 18/48 | 18/49
Serious Adverse Events (participants affected / at risk) | 4/48 | 14/49
Other Adverse Events (participants affected / at risk) | 43/48 | 44/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium 223 Dichloride (N=48) | Placebo (N=49)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (2)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium 223 Dichloride (N=48) | Placebo (N=49)
Anaemia (Blood and lymphatic system disorders) | 3 (5) | 3 (7)
Leukopenia (Blood and lymphatic system disorders) | 3 (6) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (12) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 2 (3)
Constipation (Gastrointestinal disorders) | 4 (5) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 10 (15) | 7 (10)
Nausea (Gastrointestinal disorders) | 12 (18) | 9 (13)
Vomiting (Gastrointestinal disorders) | 7 (7) | 7 (11)
Fatigue (General disorders) | 12 (15) | 9 (10)
Influenza like illness (General disorders) | 3 (4) | 1 (1)
Oedema peripheral (General disorders) | 3 (3) | 1 (1)
Pain (General disorders) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 4 (5)
Traumatic fracture (Injury, poisoning and procedural complications) | 2 (3) | 4 (6)
Weight decreased (Investigations) | 3 (5) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (14) | 11 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (18) | 7 (10)
Bone pain (Musculoskeletal and connective tissue disorders) | 11 (12) | 9 (15)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (10) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (8) | 7 (9)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 6 (8) | 7 (8)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (3)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (7)
Dizziness (Nervous system disorders) | 2 (3) | 3 (3)
Headache (Nervous system disorders) | 13 (19) | 4 (4)
Paraesthesia (Nervous system disorders) | 1 (1) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Hypertension (Vascular disorders) | 3 (5) | 3 (5)
Hot flush (Vascular disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
Due to the premature enrollment discontinuation, reduced sample size, and potentially curtailed active follow up, the planned number of SSE FS events was not achieved, limiting the assessment of the primary efficacy endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT02258464/SAP_000.pdf
  • Study Protocol (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT02258464/Prot_001.pdf